CLINICAL TRIAL: NCT07047417
Title: Confocal Laser Endomicroscopy Combined With Rapid On-Site Cytological Evaluation for the Diagnosis of Intrathoracic Lymphadenopathy
Brief Title: Optical Biopsy and Cytological Evaluation for Intrathoracic Lymphadenopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Director, Department of Respiratory Endoscopy, Shanghai Chest Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KS25034
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Intrathoracic Lymphadenopathy
Keywords: confocal laser endomicroscopy; rapid on-site evaluation; intrathoracic lymphadenopathy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with intrathoracic lymphadenopathy (Experimental): Approximately 150 patients with intrathoracic lymphadenopathy who meet the inclusion and exclusion criteria will be prospectively included. CLE and ROSE will be performed to diagnose the lesion. 100 patients will be used to establish CLE and ROSE interpretation criteria, and 50 patients will be used for criteria validation.
  Interventions: Diagnostic Test: CLE and ROSE

INTERVENTIONS:
Diagnostic Test: CLE and ROSE — All patients undergo white light bronchoscopy after general anesthesia to rule out abnormalities in the lumen and clear the airways. After locating the target lymph node using convex probe endobronchial ultrasound (CP-EBUS), the target lymph node is routinely explored using the grayscale, blood flow and elastography modes CP-EBUS. Puncture is performed using a puncture needle under the guidance of CP-EBUS, and then the CLE probe is inserted into the target lymph node through the puncture needle. Sodium fluorescein is intravenously injected before CLE imaging. Under the guidance of CP-EBUS, the CLE probe is slowly moved to examine the target lesion. According to the real-time CLE images, the ideal biopsy location is identified. After the CLE examination is completed, cryobiopsy is performed at the ideal biopsy location confirmed by CLE under the guidance of CP-EBUS. After sampling, ROSE of the samples is performed.

SUMMARY:
The purpose of this study is to describe and validate confocal laser endomicroscopy(CLE) and rapid on-site evaluation(ROSE) interpretation criteria for different types of intrathoracic lymphadenopathy.

DETAILED DESCRIPTION:
This is a single-arm, single-center and prospective study. Approximately 150 patients with intrathoracic lymphadenopathy will be included to receive CLE and ROSE for the diagnosis of the lesions. CLE is a modern imaging technique that uses an excitation laser light to create real-time microscopic images of tissues. During transbronchial biopsy, CLE has the potential to provide rea-lime non-invasive diagnosis of intrathoracic lymphadenopathy ('optical biopsy'). Rapid on-site evaluation (ROSE) is an important auxiliary technology for transbronchial biopsy, providing rapid cytopathological evaluation of specimens during operation and feedback on specimen quality and preliminary diagnosis of lesions. In this study, we will obtain CLE images and ROSE images of the target lesion . We will compare the results of the 'optical biopsy' and cytological evaluation with the corresponding histopathological results and develop CLE and ROSE interpretation criteria for different types of intrathoracic lymphadenopathy. In addition, we will perform the validation of these criteria to evaluate the ability of CLE and ROSE to discriminate between benign and malignant intrathoracic lymphadenopathy.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old.
2. Chest CT shows at least one enlarged intrathoracic lymph node (short axis >1 cm), or PET / CT shows increased fluorodeoxyglucose uptake (standard uptake value > 2.5) in at least one intrathoracic lymph node.
3. CP-EBUS-TBNA is required to determine the diagnosis or staging.
4. Patients who have good compliance and sign informed consent.

Exclusion Criteria:

1. Patients with known allergy for fluorescein.
2. Pregnant or lactating women.
3. Patients with contraindications of bronchoscopy.
4. The investigators believe that patient has other conditions that are not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of CLE combined with ROSE in differential diagnosis of benign and malignant intrathoracic lymphadenopathy | 6 month post-procedure
  Diagnostic accuracy is defined as the number of lesions correctly identified as malignant or benign using our proposed CLE and ROSE interpretation criteria divided by the total number of lesions.

SECONDARY OUTCOMES:
Sensitivity, specificity, positive predictive value and negative predictive value of CLE combined with ROSE in differential diagnosis of benign and malignant intrathoracic lymphadenopathy | 6 months post-procedure
  Sensitivity is defined as the number of lesions correctly identified as malignant using our proposed CLE and ROSE interpretation criteria divided by the total number of malignant lesions. Specificity is defined as the number of lesions correctly identified as benign using our proposed CLE and ROSE interpretation criteria divided by the total number of benign lesions. The positive predictive value is the percentage of true malignant lesions among all lesions identified as malignant using our proposed CLE and ROSE interpretation criteria. The negative predictive value is the percentage of true benign lesions among all lesions identified as benign using our proposed CLE and ROSE interpretation criteria.
Accuracy, sensitivity, specificity, positive predictive value and negative predictive value of CLE alone in differential diagnosis of benign and malignant intrathoracic lymphadenopathy | 6 months post-procedure
  Accuracy is defined as the number of lesions correctly identified as malignant or benign using our proposed CLE interpretation criteria divided by the total number of lesions. Sensitivity is defined as the number of lesions correctly identified as malignant using our proposed CLE interpretation criteria divided by the total number of malignant lesions. Specificity is defined as the number of lesions correctly identified as benign using our proposed CLE interpretation criteria divided by the total number of benign lesions. The positive predictive value is the percentage of true malignant lesions among all lesions identified as malignant using our proposed CLE interpretation criteria. The negative predictive value is the percentage of true benign lesions among all lesions identified as benign using our proposed CLE interpretation criteria.
Accuracy, sensitivity, specificity, positive predictive value and negative predictive value of ROSE alone in differential diagnosis of benign and malignant intrathoracic lymphadenopathy | 6 months post-procedure
  Accuracy is defined as the number of lesions correctly identified as malignant or benign using our proposed ROSE interpretation criteria divided by the total number of lesions. Sensitivity is defined as the number of lesions correctly identified as malignant using our proposed ROSE interpretation criteria divided by the total number of malignant lesions. Specificity is defined as the number of lesions correctly identified as benign using our proposed ROSE interpretation criteria divided by the total number of benign lesions. The positive predictive value is the percentage of true malignant lesions among all lesions identified as malignant using our proposed ROSE interpretation criteria. The negative predictive value is the percentage of true benign lesions among all lesions identified as benign using our proposed ROSE interpretation criteria.
Diagnosis accuracy of CLE combined with ROSE in differential diagnosis of different types of intrathoracic lymphadenopathy | 6 months post-procedure
  Different types of common malignant intrathoracic lymphadenopathy include pulmonary adenocarcinoma, squamous cell lung carcinoma, small cell lung carcinoma and so on. Different types of common benign intrathoracic lymphadenopathy include tuberculosis, sarcoidosis, fungal infection and so on.
Diagnosis accuracy of CLE or ROSE alone in differential diagnosis of different types of intrathoracic lymphadenopathy | 6 months post-procedure
  Different types of common malignant intrathoracic lymphadenopathy include pulmonary adenocarcinoma, squamous cell lung carcinoma, small cell lung carcinoma and so on. Different types of common benign intrathoracic lymphadenopathy include tuberculosis, sarcoidosis, fungal infection and so on.
Incidence of complications | 1 month post-procedure
  Complications mean a composite of procedure related adverse advents during and after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Jiayuan Sun, Study Director — Shanghai Chest Hospital
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No